CLINICAL TRIAL: NCT03495336
Title: A 4-week Consumption of Light or Dark Roast Unfiltered (Turkish) Coffee Affects Cardiovascular Risk Parameters of Homocysteine and Cholesterol Concentrations in Healthy Subjects: A Randomized Crossover Clinical Trial
Brief Title: The Effects of Unfiltered (Turkish) Coffee Consumption on Cardiovascular Risk Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Fatma Hülyam Eren, Instructor, Eastern Mediterranean University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: EasternMedU
Record Dates: First submitted 2018-03-17; First posted 2018-04-12 (Actual); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Cardiovascular Diseases
Keywords: Boiled coffee; Cardiovascular disease; Cholesterol; Homocysteine; Turkish coffee; Diterpenes; Unfiltered coffee
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Washout period (Experimental): Coffee abstention phase for 2 weeks.
  Interventions: Other: coffee abstention phase
- Light roast coffee (LR) (Experimental): Participants will follow LR Coffee consumption procedure and consume at least 3 cups of Light (LR) roast Turkish coffee brews per day for 4 weeks after a washout period (WO) of 2 weeks.
  Interventions: Other: LR Coffee consumption
- Second washout period (Experimental): coffee abstention phase for 2 weeks
  Interventions: Other: coffee abstention phase
- Dark roast coffee (DR) (Experimental): Participants will follow DR Coffee consumption procedure and consume at least 3 cups of Dark (DR) roast Turkish coffee brews per day for 4 weeks after a washout period (WO) of 2 weeks.
  Interventions: Other: DR Coffee consumption

INTERVENTIONS:
Other: coffee abstention phase — no coffee consumption for 2 weeks
  Arms: Second washout period; Washout period
Other: LR Coffee consumption — for 4 weeks participants consumed only LR Turkish coffee
  Arms: Light roast coffee (LR)
Other: DR Coffee consumption — for 4 weeks participants consumed only DR Turkish coffee
  Arms: Dark roast coffee (DR)

SUMMARY:
Purpose/Objective: The aim of this study is to investigate the impact of boiled unfiltered (Turkish) coffee consumption on the plasma cardiovascular risk parameters of healthy subjects. The study also explores whether two unfiltered boiled (Turkish) coffee beverages that differ in content due to different roasting degrees will differentially affect cardiovascular biomarkers.

Methods: In this crossover intervention study, healthy, nonsmoking, habitual Turkish coffee drinkers (n=28) were randomized to consume at least 3 cups of Light (LR) or Dark (DR) roast Turkish coffee brews per day for 4 weeks after a washout period (WO) of 2 weeks. Subsequent to each coffee abstinence period, both groups received the alternative intervention. After the first WO and the coffee intervention periods, anthropometric measures, blood pressure, heart rate and 13 biochemical parameters were collected and dietary records were completed.

DETAILED DESCRIPTION:
Background: Considerable controversy exists regarding the link between coffee consumption and cardiovascular disease (CVD) risk. It has been shown that different coffee preparation and brewing methods influence the concentration of compounds present in the final coffee brew. Unlike coffee traditionally consumed in the western world, Turkish coffee is not drip filtered, but rather its method of preparation involves slowly boiling water that is mixed with thinly ground coffee beans. This style of preparation results in a greater amount of biologically active components (caffeine and diterpenes) remaining in the liquid. In addition to preparation styles, roasting process greatly affects the chemical composition of the coffee. Coffee types differing in content of major constituents differ with regard to cardiovascular health effects.

Purpose/Objective: The aim of this study is to investigate the impact of boiled unfiltered (Turkish) coffee consumption on the plasma cardiovascular risk parameters of healthy subjects. The study also explores whether two unfiltered boiled (Turkish) coffee beverages that differ in content due to different roasting degrees will differentially affect cardiovascular biomarkers.

Methods: In this crossover intervention study, healthy, nonsmoking, habitual Turkish coffee drinkers (n=28) were randomized to consume at least 3 cups of Light (LR) or Dark (DR) roast Turkish coffee brews per day for 4 weeks after a washout period (WO) of 2 weeks. Subsequent to each coffee abstinence period, both groups received the alternative intervention. After the first WO and the coffee intervention periods, anthropometric measures, blood pressure, heart rate and 13 biochemical parameters were collected and dietary records were completed.

ELIGIBILITY:
Inclusion Criteria:

* Regular Turkish coffee consumer ≥ 1 cups/day
* Body mass index (BMI) 18.5-24.9 kg/m2 )
* Non-smoker or former smoker (more than a year)
* Willingness to abstain from coffee drinking
* Willingness to consume ≥ 3 cups/day of Turkish coffee

Exclusion Criteria:

* Acute or chronic diseases
* Severe illness with in-patient treatment during last 3 months
* Use of regular medication or any supplements
* Weight reduction ˃2 kg/week during the last month
* Pregnancy or breastfeeding
* Regular strong physical activity with ≥1h/day
* High alcohol intake a weekly intake of ˃7 units for women and ˃14units for men
* Excess consumption of total fat ˃35% of daily calories
* Consumption of saturated fatty acid ˃10% of daily calories
* Cholesterol intake ˃300mg/day

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2017-06-22 (Actual); Study Completion 2017-10-22 (Actual)

PRIMARY OUTCOMES:
Comparing the serum lipid levels of all interventions | 12 weeks
  Differences in concentration of serum lipid levels of participants in coffee-free period (washout) and after LR or DR coffee ingestion were measured.
  Blood samples were obtained at the end of two weeks washout period and after each four weeks coffee intervention period, and sera were stored at -30∘ C, until analytical measurements were performed. The levels of serum lipids: Triglycerides (mg/dL), Total cholesterol (mg/dL), and HDL cholesterol (mg/dL) were determined using a Dimension Xpand Plus integrated clinical chemistry autoanalyzer (Siemens Healthcare Diagnostics, Deerfield, IL, USA). The serum levels of LDL cholesterol (mg/dL) were calculated using Friedewald's equation. Differences in blood lipid variables were analyzed by repeated-measures ANOVA for comparisons of LR coffee intake with DR and of each roast with the washout.analyses were performed using SPSS 24.0 (IBM-SPSS Inc., Chicago, IL, USA).

SECONDARY OUTCOMES:
Comparing the weight (kg) of all interventions | 12 weeks
  Weight was measured after the washout period and after each intervention. Weight (in kilograms) was measured in light clothing, without shoes.
Comparing the height (cm) of all interventions | 12 weeks
  after the washout period and after each intervention height was measured using a stadiometer to the nearest centimeter.
Comparing the body mass index (BMI) of all interventions | 12 weeks
  BMI was calculated (weight/height squared; in kilograms per square meter)
Comparing the body fat percentage (%) of all interventions | 12 weeks
  after the washout period and after each intervention the percentage of body fat and fat free mass (FFM) was measured by Tanita Segmental Body Composition Analyzer BC-418 MA (Tanita Corp. Tokyo, Japan)
Comparing the waist circumference (cm) of all interventions | 12 weeks
  after the washout period and after each intervention waist circumferences (midway between the rib cage and the iliac crest) were measured using a flexible tape.
Comparing the blood pressure (BP) (Systolic and Diastolic blood pressure (mmHg)) of all interventions | 12 weeks
  after the washout period and after each intervention BP and heart rate (beats/min) was monitored using an automatic arm sphygmomanometer (Pic Indolor Diagnostic, BS 150, Artsana, Italy) after a 5-min rest in a sitting position.
Comparing the 3-day food diaries (1 weekend day and 2 weekdays) taken during each intervention | 12 weeks
  Daily nutrient intake was calculated by using computer software (Ebispro, Stuttgart, Germany; Turkish version: BeBiS, Vers. 6.1)
Comparing the physical activity levels of each intervention | 12 weeks
  The validated Turkish version of the International Physical Activity Questionnaire (IPAQ)-short form (7 item) was administered. The IPAQ questionnaires list activities and request estimates of durations and frequencies for each activity engaged in over the past week. Durations are multiplied by known METs per activity and the results for all items are summed for the overall physical activity score. Scores for walking and for moderate and vigorous activities are sums of corresponding item scores. A sitting question is not included in physical activity score. Physical activity level (PAL): Extremely inactive <1.40 , Sedentary 1.40-1.69, Moderately active 1.70-1.99, Vigorously active 2.00-2.40,Extremely active>2.40
Comparing the Homocysteine levels of all interventions | 12 weeks
  Differences in concentration of homocysteine (μmol/L) levels of participants after 2wk coffee-free period (washout) and after 4 weeks of LR or DR coffee ingestion was compared. EDTA-treated blood samples for total homocysteine (μmol/L) analysis were immediately refrigerated (placed on ice) until the plasma was separated by centrifugation. All the samples were assayed for Homocysteine by using High Performance Liquid Chromatography with fluorescent detection technique (HPLC-FLD). Differences in homocysteine variables were analyzed by repeated-measures ANOVA for comparisons of LR coffee intake with DR and of each roast with the washout.analyses were performed using SPSS 24.0 (IBM-SPSS Inc., Chicago, IL, USA).
Comparing the fasting blood glucose levels of all interventions | 12 weeks
  Concentration of fasting blood glucose levels in coffee-free period (washout) and changes after LR or DR coffee ingestion were compared.Blood samples were obtained at the end of two weeks washout period and after each four weeks coffee intervention period, and sera were stored at -30∘ C, until analytical measurements were performed. The levels of Fasting blood glucose (mg/dL), were determined using a Dimension Xpand Plus integrated clinical chemistry autoanalyzer (Siemens Healthcare Diagnostics, Deerfield, IL, USA). Differences in human variables were analyzed by repeated-measures ANOVA for comparisons of LR coffee intake with DR and of each roast with the washout.
Comparing the serum Malondialdehyde levels of all interventions | 12 weeks
  Concentration of Serum Malondialdehyde (μM) levels at the end of coffee-free period (washout) and changes after LR or DR coffee ingestion were compared.Serum Malondialdehyde (μM) levels were determined with a colorimetric assay kit (Cayman Chemical, Ann Arbor, MI). Differences in human variables were analyzed by repeated-measures ANOVA for comparisons of LR coffee intake with DR and of each roast with the washout.

OTHER OUTCOMES:
Analysis of the content of the diterpenes (cafestol and kahweol) (mg/55mL) in LR and DR Turkish coffee brews | 3 months
  Cafestol and kahweol were analyzed in the unsaponified matter by HPLC-DAD. Diterpenes content of the two coffee beverages were reported as mean±standard deviation and Kruskal-Wallis test was used for statistical comparison of coffee roasts.. All analyses were performed using SPSS 24.0 (IBM-SPSS Inc., Chicago, IL, USA).
Analysis of the content of the caffeine (mg/mL) in LR and DR Turkish coffee brews | 3 months
  Caffeine was determined by high-performance liquid chromatography (HPLC, Aligent Technologies, USA) with diode-array detector (DAD) and mass spectrometer. content of the two coffee beverages were reported as mean±standard deviation and Kruskal-Wallis test was used for statistical comparison of coffee roasts.. All analyses were performed using SPSS 24.0 (IBM-SPSS Inc., Chicago, IL, USA).

CONTACTS AND LOCATIONS:
Overall Officials: Tanju Besler, Prof., Study Chair — Eastern Mediterranean University
Locations (1):
- Eastern Mediterrenean University, Famagusta, Cyprus

IPD SHARING:
Plan to Share IPD: Undecided